CLINICAL TRIAL: NCT01824927
Title: Pain Expression in the Perioperative Period of Cataract Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Evidence Based Cataract Study Group (Other)
Responsible Party: Principal Investigator, Peng ZHOU, Secretary of EBCS Group, Evidence Based Cataract Study Group
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: EBCS001; NSFC81200669 (Other Grant/Funding Number: National Natural Science Foundation of China (NSFC, No. 81200669))
Record Dates: First submitted 2013-04-02; First posted 2013-04-05 (Estimated); Last update posted 2013-04-05 (Estimated); Status verified 2013-04

CONDITIONS: Cataract; Surgery; Eye Pain
MeSH Terms: conditions — Cataract; Eye Pain

STUDY DESIGN:
Who Masked: Participant

ARMS (3):
- First eye (FE) (Active Comparator): Phacoemulsification cataract extraction surgery of first eye
  Interventions: Procedure: First eye (FE); Drug: Steroids eye drops
- Second eye (SE) (Active Comparator): Phacoemulsification cataract extraction surgery of second eye
  Interventions: Procedure: Second eye (SE); Drug: Steroids eye drops
- Steroids eye drops (Experimental): Dexamethasone eye drop, 1 drop, qid, for 3 days before surgery
  Interventions: Procedure: First eye (FE); Procedure: Second eye (SE)

INTERVENTIONS:
Procedure: First eye (FE) — Phacoemulsification cataract extraction surgery
  Arms: First eye (FE); Steroids eye drops
Procedure: Second eye (SE) — Phacoemulsification cataract extraction surgery
  Arms: Second eye (SE); Steroids eye drops
Drug: Steroids eye drops — Use steroids eye drops to decrease the pain.
  Arms: First eye (FE); Second eye (SE)

SUMMARY:
Patients having cataract extraction in the second eye under topical anesthesia with monitored anesthesia care often report increased pain and awareness relative to the first surgery in the fellow eye, despite similar operative and anesthetic conditions. The purpose of this study is to investigate the pathogenesis of this phenomenon.

ELIGIBILITY:
Inclusion Criteria:

* Age-related cataract patients aged 50 years or older able to give informed consent undergoing cataract surgery;
* Pupil dilation ≧7 mm after mydrisis;
* VA prognosis ≧6/12

Exclusion Criteria:

* Unable to give informed consent;
* Patients with history of ocular pathology or diabetic retinopathy;
* Patients with traumatic, subluxated and posterior polar cataract;
* Patients had other ocular surgery (not cataract surgery) in the past 6 months;
* Patients with significant intra-operative complications

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2013-01; Primary Completion 2013-05 (Estimated)

PRIMARY OUTCOMES:
Post operative pain level | 3 days
  Post operative pain level recorded on a VAS (0-10) at rest for the first three days after cataract surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Eye and ENT Hospital of Fudan University, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Zhu XJ, Wolff D, Zhang KK, He WW, Sun XH, Lu Y, Zhou P. Molecular Inflammation in the Contralateral Eye After Cataract Surgery in the First Eye. Invest Ophthalmol Vis Sci. 2015 Aug;56(9):5566-73. doi: 10.1167/iovs.15-16531. PMID 26305528